CLINICAL TRIAL: NCT04562025
Title: Clinical Research of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSCs) in the Treatment of Diabetic Nephropathy
Brief Title: Clinical Research of UC-MSCs in the Treatment of Diabetic Nephropathy
Acronym: UC-MSCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Wuhan Hamilton Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200915HMD
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy; Safety; Efficiency; Cell Therapy; UC-MSCs
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-MSCs treatment group (Experimental): Conventional treatment plus UC-MSCs:
  Participants will receive conventional treatment plus 3 times of UC-MSCs (1*10E6 UC-MSCs/kg body weight/100mL intravenously at week 1, week 2，week3).
  Interventions: Drug: UC-MSCs
- Placebo control group (Placebo Comparator): Conventional treatment plus Placebo:
  Without UC-MSCs therapy but conventional treatment should be received. Participants will receive conventional treatment plus 3 times of Placebo intravenously at week 1, week 2，week3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UC-MSCs — 3 times of UC-MSCs (1*10E6 UC-MSCs/kg body weight/100mL saline containing 1% human albumin intravenously at week 1,week 2, week 3).
  Other Names: UC-MSCs treatment group
  Arms: UC-MSCs treatment group
Drug: Placebo — 3 times of cell-free stem cell suspension (saline containing 1% human albumin/100mL intravenously at week 1, week 2, week 3).
  Other Names: Placebo control group
  Arms: Placebo control group

SUMMARY:
Diabetic nephropathy (DN) is one of the most serious complications of diabetes and the leading cause of end-stage chronic kidney disease. DN is a refractory disease with low awareness, high incidence, and high disability. The incidence of DN can reach 30 to 40% after 20 years of diabetes, of which 5~10% of patients will progress to end-stage renal disease, and epidemiological surveys predict that by 2030, DN will become the seventh leading cause of death in the world. Currently, there are no effective drugs for treating DN. This clinical trial is to inspect the safety and efficiency of human umbilical cord mesenchymal stem cells (UC-MSCs) therapy for patients with DN.

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is one of the most important microvascular complications of diabetes. It is a persistent and refractory disease. There is currently a lack of effective clinical treatments for DN. The basic pathological processes of DN are renal tissue cell damage, apoptosis and continuous increase of inflammatory cytokines induced by early high glucose, which gradually leads to glomerular sclerosis and renal fibrosis.

Human umbilical cord mesenchymal stem cells (UC-MSCs), as the "youngest" adult stem cells, have powerful anti-inflammatory functions, stronger differentiation potential, and good safety. They are ideal seed cells for the treatment of DN. At present, studies on a variety of animal models of DN have shown that mesenchymal stem cell transplantation can delay the progression of DN and have a certain repair effect on damaged kidney tissue and renal function. Our previous preclinical study showed that UC-MSCs effectively improved the renal function, inhibited inflammation and fibrosis, and prevented its progression in a rat model of diabetes-induced chronic renal injury. Some autologous or allogeneic mesenchymal stem cells have been carried out abroad treatment of chronic kidney disease caused by various reasons, including clinical trials of DN, phase I/II test results did not show obvious adverse reactions related to stem cell therapy, and can improve the patient's renal function and quality of life to a certain extent.

The purpose of this study is to investigate efficiency and safety of UC-MSCs in treating DN patients. This trial will recruit 38 patients. 19 patients received the treatment of conventional treatment + equal volume normal saline containing 1% human albumin (placebo group) were used as control group; conventional treatment + 1*10E6 UC-MSCs/kg body weight (experimental group) for intravenous infusion (once a week, 3 times in total) to treat 19 patients with DN (by unified standard inclusion), and subjects will be followed a total of 48 weeks from time of initial cell treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus, course 5-15 years;
2. Age 30-65 years old, no gender limit;
3. Accompanied by proteinuria, urine albumin/creatinine ratio (UACR)>300mg/g or 24h urine protein quantitative>0.5g/24h;
4. eGFR is between 30-60 ml/min/1.732 m2;
5. Take RASI-based antihypertensive drugs to control blood pressure and blood pressure meets the following standards: systolic blood pressure <150mmHg, and diastolic blood pressure <100mmHg;
6. Blood lipids and blood uric acid are controlled at appropriate levels;
7. The pathological diagnosis of kidney biopsy is diabetic nephropathy;
8. Patients who have good compliance, signed informed consent, and can complete the entire trial treatment and follow-up plan according to the research plan；
9. No exclusion criteria are positive.

Exclusion Criteria:

1. Have a history of primary glomerulonephritis, lupus nephritis, ANCA-related small vasculitis, renal damage, allergic purpura nephritis, hepatitis B-related nephritis;
2. Poor blood glucose control: HbA1c ≥9% of patients or 2h postprandial blood glucose> 22mmol/L;
3. Active liver disease or liver function test results are obviously abnormal (ALT or AST ≥ 2 times the upper limit of normal);
4. White blood cell count<3.0×10E9/L, hemoglobin<80 g/L, platelet count<100×10E9/L or suffering from other blood system diseases (severe anemia, idiopathic thrombocytopenic purpura, splenomegaly, Patients with coagulopathy, etc.);
5. Severe and unstable cardiovascular and cerebrovascular diseases (unstable angina pectoris, coronary artery disease, cerebrovascular disease, transient ischemic attack, congestive heart failure, etc.), acute and uncontrollable disease, still unable to effectively control severe hypertension (blood pressure> 160/100 mmHg) after treatment or organ transplant patients;
6. The dose of antihypertensive drugs and/or hypoglycemic drugs used in the past 3 months has increased significantly than before;
7. Uncontrolled infection;
8. Suffer from tumor or abnormal level of tumor markers;
9. Suffer from blood-borne diseases (for example, HIV, syphilis, hepatitis B and hepatitis C);
10. Possibility of pregnancy, preparation for pregnancy or breastfeeding;
11. Receive immunosuppressive treatment;
12. Have a history of allergies, especially those who are allergic to human albumin;
13. Suffer from mental illness, which will affect their voluntariness, decision-making ability and communication ability;
14. A history of alcohol abuse or a known history of drug abuse in the last 2 years;
15. Participate in another clinical trial within the last 3 months;
16. Poor compliance, unable to complete the entire study；
17. The researcher diagnosed that the patient is not suitable for this study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From Baseline (0 W) to 48 weeks after treatment
  The number of Adverse Events associated with UC-MSCs intervention per treatment arm
Adverse Events | From Baseline (0 W) to 48 weeks after treatment
  The percentage of Adverse Events associated with UC-MSCs intervention per treatment arm

SECONDARY OUTCOMES:
Kidney function | From Baseline (0 W) to 48 weeks after treatment
  Change in estimated glomerular filtration rate (eGFR) from baseline.
Kidney function | From Baseline (0 W) to 48 weeks after treatment
  Change in 24-hour urinary protein quantification from baseline.
Kidney function | From Baseline (0 W) to 48 weeks after treatment
  Change in urinary albumin/creatinine ratio from baseline
Kidney function | From Baseline (0 W) to 48 weeks after treatment
  The proportion of subjects in both groups who progressed to end-stage renal disease (ESRD) or doubled their serum creatinine.
SF-36 (The MOS item short from health survey) | From Baseline (0 W) to 48 weeks after treatment
  The MOS item short from health survey, SF-36 and changes per visit. As a concise health questionnaire, SF-36 comprehensively summarizes the quality of life of the surveyed from 8 aspects: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. Higher scores mean a better outcome.
Change in HbA1c | From Baseline (0 W) to 48 weeks after treatment
  Change in Glycosylated Hemoglobin (HbA1c) from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan university, Wuhan, Hubei China, China